CLINICAL TRIAL: NCT01818856
Title: Pharmacokinetic Interactions Between Telaprevir and Un-boosted Atazanavir in HIV/HCV-co-infected Patients Under Treatment for Genotype 1 Chronic Hepatitis C.
Brief Title: Pharmacokinetic Interactions Between Telaprevir and Un-boosted Atazanavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Luis F. Lopez-Cortes, MD, PhD, Hospitales Universitarios Virgen del Rocío
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LLC-TEL-2012-1; 2012-002515-25 (EudraCT Number)
Record Dates: First submitted 2012-12-29; First posted 2013-03-27 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Hepatitis C, Chronic; HIV Infection
Keywords: Chronic hepatitis C; HIV-infection; Drug interaction
MeSH Terms: conditions — Hepatitis C, Chronic; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Telaprevir interactions (Experimental): Telaprevir 750 mg/8h or 1125 mg/12h (+ pegIFN alfa and ribavirin) plus Atazanavir/ritonavir 300/100 mg/24. Pharmacokinetic profile on day 0.
  Intervention: Ritonavir will be withdrawn and the atazanavir dose increased to 200 mg/12h for days 1 to 7. On day 8: a morning dose of Telaprevir (750 mg or 1125 mg) plus Atazanavir 200 mg. Pharmacokinetic profile for 12 hours
  Interventions: Drug: Ritonavir withdrawal, atazanavir 200 mg/12h; Drug: Telaprevir interactions

INTERVENTIONS:
Drug: Ritonavir withdrawal, atazanavir 200 mg/12h
  Other Names: Reyataz; Norvir; Incivo
Drug: Telaprevir interactions
  Other Names: Incivo; Reyataz; Norvir

SUMMARY:
Hypothesis: the Telaprevir(TVR) plasma levels (750 mg q8h or 1125 mg/12h )will not be affected when co-administered with un-boosted Atazanavir (ATV) 200 mg q12h plus two analogues (NRTIs) in HCV/HIV-co-infected patients.

DETAILED DESCRIPTION:
Objectives

1. Primary Outcome Measures: evaluate the changes in the plasma pharmacokinetic parameters (Cmax, Cmin, AUC, t 1/2, and Cl) of Telaprevir (TVR) administered at 750 mg/8h together with un-boosted Atazanavir (200 mg/12h), taking as reference the pharmacokinetic parameters observed when TVR is administered with Atazanavir/ritonavir (300/100 mg/day)
2. To assess the changes in the plasma pharmacokinetic parameters of Atazanavir administered as 200 mg/12h with respect to its administration as 300/100 mg/day when administered together with TVR (750 mg/8h or 1125 mh/12h).

Method: open labelled clinical trial with a planned duration of 24 weeks in which 14 HIV/Hepatitis C virus genotype 1 patients under treatment with pegylated α-interferon, Ribavirin and Telaprevir will be enrolled. A 24 hours pharmacokinetic profile will be obtained after a supervised drug intake while taking TVR and ATV/rtv. Afterwards, the patients will take un-boosted ATV 200 mg bid for 7 - 10 days. Subsequently, a new pharmacokinetic profile will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old co-infected with HIV and genotype 1 HCV under treatment with pegylated α-interferon, Ribavirin and Telaprevir according to the recommendations of the Spanish Agency of Medicines and Health Products.
* Informed consent of the patient.

Exclusion Criteria:

* The usual exclusion criteria in clinical practice to start the treatment with these drugs (pegylated α-interferon, Ribavirin, Telaprevir and atazanavir) according to the Spanish and international recommendations (Spanish Agency of Medicines and Health Products,European Association for the Study of the Liver Clinical Practice Guidelines: management of hepatitis C virus infection. J Hepatol. 2011. Consensus Document of Gesida/Spanish Plan on Aids regarding the antiretroviral treatment in adults infected with the human immunodeficiency virus [Updated January 2012]).
* Concomitant use of drugs or medicinal products that could alter the pharmacokinetics of TVR or ATV.
* Medical records suggesting malabsorption or presence of diarrhea (>3 depositions/day) that could interfere with the absorption of the studied drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Changes in pharmacokinetic parameters of TVR | 7 - 10 days
  The Telaprevir peak concentrations (Cmax), trough levels (Cmin) at 8 or 12 hours, the areas under the curves over the dosing interval (AUC0-τ), and half-life during the elimination phase (t½ β) will be compared between days 0 and 7 as geometric mean ratios (GMRs) and their 90% CIs using day 0 values as reference. The differences in pharmacokinetic parameters between the regimens will be considered significant when the interval between low and high 90% CI did not include the value 1.0.

SECONDARY OUTCOMES:
Changes in pharmacokinetic parameters of ATV | 7 - 10 days
  The Atazanavir peak concentrations (Cmax), trough levels (Cmin) at 12 or 24 hours, the areas under the curves over the dosing interval (AUC0-τ), and half-life during the elimination phase (t½ β) will be summarized as geometric means (GM) and will be compared between days 0 and 7 as geometric mean ratios (GMRs) and their 90% CIs using day 0 values as reference. The differences in pharmacokinetic parameters between the regimens will be considered significant when the interval between low and high 90% CI did not include the value 1.0.

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Lopez-Cortes, MD, PhD., Principal Investigator — Instituto de Biomedicina de Sevilla (IBiS), Hospital Universitario Virgen del Rocío/CSIC/Universidad de Sevilla. Spain.
Locations (1):
- Hospital Universitario Virgen del Rocio, Seville, Seville, Spain

REFERENCES:
- [Derived] Gutierrez-Valencia A, Ruiz-Valderas R, Ben-Marzouk-Hidalgo OJ, Torres-Cornejo A, Espinosa N, Castillo-Ferrando JR, Viciana P, Lopez-Cortes LF. Telaprevir and ribavirin interaction: higher ribavirin levels are not only due to renal dysfunction during triple therapy. Antimicrob Agents Chemother. 2015;59(6):3257-62. doi: 10.1128/AAC.04795-14. Epub 2015 Mar 23. PMID 25801562
- [Derived] Gutierrez-Valencia A, Ruiz-Valderas R, Torres-Cornejo A, Viciana P, Espinosa N, Castillo-Ferrando JR, Lopez-Cortes LF. Role of ritonavir in the drug interactions between telaprevir and ritonavir-boosted atazanavir. Clin Infect Dis. 2014 Jan;58(2):268-73. doi: 10.1093/cid/cit693. Epub 2013 Oct 21. PMID 24145880